CLINICAL TRIAL: NCT03207230
Title: A Multicenter Exploratory Study of Accelerometry Measurements in Dilated Cardiomyopathy Patients
Brief Title: Multicenter Exploratory Study of Accelerometry in Dilated Cardiomyopathy
Acronym: MESA-DCM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding not secured
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Matthew Wheeler, Clinical Assistant Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 41695
Record Dates: First submitted 2017-06-27; First posted 2017-07-02 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Dilated Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Intervention Model Description: All participants enrolled in the study will receive the wearables and will be evaluated for the relationship between daily physical activity levels and functional capacity (VO2 peak).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Standard (Experimental): All participants will perform the CPET at Baseline visit and will be provided with the Cardea SOLO, ActiGraph wGT3X-BT and Wavelet Wristband. The participants will be asked to response to KCCQ and Stanford 7 day recall surveys.
  Interventions: Device: Cardea SOLO; Device: ActiGraph wGT3X-BT; Device: Wavelet Wristband

INTERVENTIONS:
Device: Cardea SOLO — Participants will be asked to wear everyday for 7 days after the Baseline visit. the monitor attaches to the skin with adhesive and records heart rate and heart rhythm.
Device: ActiGraph wGT3X-BT — Participants will be asked to wear everyday for 2 weeks after the Baseline visit. The wearable tracks activity and the step count during the day.
Device: Wavelet Wristband — Participants will be asked to wear everyday for 2 weeks after the Baseline visit. The wearable measures the activity and the heart rate as measured by PPG sensor.

SUMMARY:
Study evaluates the relationships between daily physical activity levels (PAL) and functional capacity (VO2peak) in patients with dilated cardiomyopathy (DCM)

DETAILED DESCRIPTION:
The study will evaluate the daily physical activity with the use of activity monitor, heart rate monitor and event monitor in patients with dilated cardiomyopathy (DCM). These wearables track the heart rate, heart rhythm, tracks activity and step count. The VO2 peak will be measured via the exercise test.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, 18-75 years of age
2. Diagnosis of dilated cardiomyopathy

   * (Unexplained left ventricular enlargement (left ventricular end diastolic dimension (LVEDD) >95th percentile for gender and height by echo or MRI)
   * (Left ventricular ejection fraction (LVEF) less than 50%)
3. CPET within 14 days prior to baseline visit with no intervening change in therapy
4. Echocardiogram or cardiac MRI within 1 year prior to baseline
5. Able to walk >100ft without limitation
6. More than 30 minutes of exercise per week for at least 3 months prior to study enrollment, and plan to continue exercising for the next two weeks (duration of study).
7. Ability to provide informed consent and willingness to complete the study (including weekly phone follow-up)

Exclusion Criteria:

1. Heart failure hospitalization within four weeks prior to enrollment
2. Non-cardiac limitation of activity

4. Prior exercise-induced syncope or exercise-induced sudden death 5. Primary exercise mode is swimming or stationary biking 6. Participation in competitive or high intensity exercise against medical advice 7. Implantable Cardiverter Defibrillator (ICD) placement in the 2 months prior to enrollment 8. Plan for surgery, device implantation, or significant change in clinical management during the two weeks of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
VO2max correlation with daily physical activity | 2 weeks
  Maximal exercise capacity as measured by Max VO2 via CPET correlation with wearable device measures of daily physical activity

SECONDARY OUTCOMES:
NYHA correlation with daily step count | 2 weeks
  Correlation between NYHA score and daily step count or maximal walking speed
KCCQ correlation with daily step count | 2 weeks
  Correlation between KCCQ score and daily step count or maximal walking speed

CONTACTS AND LOCATIONS:
Overall Officials: Matthew T Wheeler, MD PhD, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: Undecided